CLINICAL TRIAL: NCT04558879
Title: The Effect of Different Exercise Modalities on Sleep Quality and Architecture in People With Parkinson's Disease
Brief Title: Exercise and Sleep in Parkinson's Disease
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Collaborators: Jewish Rehabilitation Hospital (Other)
Responsible Party: Principal Investigator, Marc Roig, Assistant Professor, McGill University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 35450
Record Dates: First submitted 2020-09-09; First posted 2020-09-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Rehabilitation; Neurosciences; Sleep; Exercise; Cardiovascular training; Resistance training; Cognition; Motor function; Quality of life
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiovascular training (Experimental): Cardiovascular training (CT) will be performed on a recumbent stepper. CT will start at low intensity, and through a linear progression will reach vigorous intensity; then, this intensity will be maintained until the end of the intervention. Each session will include five minutes of warm-up and cool-down performed at the beginning and the end of the training, respectively. Furthermore, five minutes of stretching will be performed after the cool down. CT's sessions will approximately last 45 minutes and will be interspersed with at least 48 hours of recovery.
  Interventions: Behavioral: CT
- Resistance training (Experimental): Resistance training (RT) intensity will be estimated using the percentage of one-maximal repetition (1-RM) defined as the maximal weight liftable for ten maximal repetitions with proper form. The program will include five exercises (leg press, lat machine, leg extension, leg curl, bench press) and will start at high-volume low-intensity. RT will follow a periodization to reach high-intensity low-volume at the end of the intervention (week 12). The training sessions will start with five-minute of warm-up performed on a recumbent stepper and will end with five-minute of stretching (cool-down). RT's sessions will approximately last 45 minutes and will be interspersed with at least 48 hours of recovery.
  Interventions: Behavioral: RT

INTERVENTIONS:
Behavioral: CT — 12 weeks of exercise Cardiovascular Training
  Arms: Cardiovascular training
Behavioral: RT — 12 weeks of exercise Resistance Training
  Arms: Resistance training

SUMMARY:
This study will investigate the impact of two common exercise modalities, cardiovascular and resistance training, on sleep quality and architecture in persons with Parkinson's disease (PD), and whether these potential positive changes in sleep are associated with improvements in brain plasticity and different quality of life (QoL)-related aspects. Participants will perform either cardiovascular training (CT) or resistance training (RT) for 12 weeks, at least two times/week. The assessments will be performed at baseline and after training by an assessor blinded to the participants' group allocation.

DETAILED DESCRIPTION:
Background: Over 100,000 Canadians are currently living with PD. Every year, 6.600 new cases are diagnosed and this number is expected to double by 2031. Most (98%) of those persons experience sleep problems, which can appear even before the onset of the cardinal motor symptoms of the disease, affecting multiple aspects of their QoL. Persons with PD also show alterations in sleep architecture, which have been associated with faster disease progression. Since medications used to reduce sleep problems in PD have potential adverse side effects, exercise has been proposed as a potential non-pharmacological alternative to improve sleep quality and architecture in people with PD. However, the most beneficial type of intervention to improve sleep in this clinical population is still to be determined.

Objective: 1) To conduct a 12-week RCT comparing the effects of CT and RT on both objective and subjective measures of sleep quality and architecture in patients with mild-to-moderate PD; 2) To assess whether, regardless of the type of exercise, positive changes in sleep quality and architecture mediate exercise-induced improvements in cognitive and motor function as well as in different aspects that directly impact on QoL; 3) To explore whether, regardless of the type of exercise used, positive changes in sleep architecture will be associated with improvements in brain plasticity and motor learning.

Design: a single-blinded RCT in which assessments will be performed at baseline (pre) and after (post) training by an assessor blinded to the participants' group allocation.

Outcomes: 1) objective and subjective sleep quality as well as sleep architecture; 2) cognitive and motor function as well as fatigue, psychological functioning, and QoL; 3) motor learning and brain plasticity.

Methods: Changes in objective (i.e. sleep efficiency) and subjective measures of sleep quality will be assessed with actigraphy and the PD sleep scale version 2, respectively. Sleep architecture will be measured with polysomnography. Motor and cognitive function will be assessed with the Unified PD Rating Scale and the Scale for Outcomes in PD-Cognition, respectively. Fatigue, psychosocial functioning and QoL will be assessed with the PD Fatigue Scale, the Scale for Outcomes in PD-Psychosocial and the PD QoL Scale, respectively. Motor learning will be assessed using a visuomotor tracking task; whereas brain plasticity will be measured with transcranial magnetic stimulation applied over the primary motor cortex.

Expected results: 1) CT will be more effective than RT in improving objective and subjective sleep quality. RT and CT will be equally effective in improving sleep architecture; 2) Improvements in sleep quality and architecture will be associated with enhancements in cognition, motor function and different QoL-related aspects; 3) Positive changes in sleep architecture will mediated increases in brain plasticity and motor learning.

Impact: This will be the first study comparing the effect of CT and RT on sleep quality and architecture and exploring associations with cognitive and motor function as well as aspects that directly impact QoL. The results of the study will provide important information to design more personalized exercise-based treatments, which are patient-oriented and aimed to mitigate sleep complains in this clinical population.

ELIGIBILITY:
Inclusion Criteria:

* Persons with mild-moderate idiopathic Parkinson's Disease (Modified Hoehn & Yahr Scale stages 1-3);
* On a stable dosage of medication during the previous month;
* Having poor sleep quality defined as a score > 18 in the PDSS-2(scores above this cut-off value define clinically relevant sleep disorders);

Exclusion Criteria:

* Having atypical parkinsonism, dementia or any other neurological, psychiatric or cardiovascular comorbidity affecting the ability to perform exercise;
* Presenting severe untreated obstructive sleep apnea (OSA);
* Having a Montreal Cognitive Assessment (MoCA) score <21
* Having a Beck Depression Inventory (BDI version 2) score >4
* Having absolute contraindications to exercise and to undergo transcranial magnetic stimulation (TMS);
* Currently are or will be enrolled in a drug or exercise trial during the duration of the study;
* Having participated in a structured exercise program > 2 times per week in the two months prior to the enrollment in the study

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency (SE) | 12 weeks
  Actigraphy; SE = total sleep time/time spent in bed.
Subjective sleep quality | 12 weeks
  Parkinson's Disease Sleep Scale version 2 (PDSS-2); Score range from 0-60; higher scores represent worse sleep quality.
Objective sleep measurements, including duration and percentage of sleep stages, total sleep time (TLT), wake after sleep onset (WASO), sleep latency (SL). | 12 weeks
  Polysomnography combined with electroencephalogram

SECONDARY OUTCOMES:
Motor function | 12 weeks
  Unified Parkinson's Disease Rating Scale part III; Scores range from 0-56; higher scores represent a worse motor function.
Cognition | 12 weeks
  Scale for Outcomes in Parkinson's Disease-Cognition; Scores range from 0-43; higher scores reflect better performance.
Fatigue | 12 weeks
  Parkinson's Disease Fatigue Scale; Scores range from 16-80; higher scores reflect a higher presence of fatigue.
Psychosocial functioning | 12 weeks
  Scale for Outcomes in Parkinson's Disease-Psychosocial; Scores range from 0-33; higher scores reflect a worse psychosocial functioning.
Quality of life-related aspects in Parkinson's disease | 12 weeks
  Parkinson's Disease Quality of Life Scale; Scores range from 0-128; higher scores indicate lower quality of life.
Motor learning | 12 weeks
  Visuomotor tracking task; accuracy in performing a novel motor task with the dominant hand.

OTHER OUTCOMES:
Intra-cortical facilitation | 12 weeks
  Paired-pulse of transcranial magnetic stimulation (TMS) protocol to estimate variation in cortical excitability measured as motor evoked potential (MEP).
Short intra-cortical inhibition | 12 weeks
  Paired-pulse of transcranial magnetic stimulation (TMS) protocol to estimate variation in cortical excitability measured as motor evoked potential (MEP).
Silent period | 12 weeks
  Paired-pulse of transcranial magnetic stimulation (TMS) protocol to estimate variation in cortical excitability measured as length of the pause in electromyographic activity.
Cardiorespiratory fitness | 12 weeks
  Maximum rate of oxygen consumption measured during maximum physical effort.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish Rehabiliation Hospital, Laval, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
Results will be published in peer-review journals.

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886